CLINICAL TRIAL: NCT05999292
Title: Phase 1 Safety and Dosimetry Study of 68Ga-R8760 in Patients With Adrenocortical Carcinoma and Healthy Volunteers
Brief Title: Phase 1 Study of 68Ga-R8760
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Radionetics Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: R8760-101
Record Dates: First submitted 2023-07-27; First posted 2023-08-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenocortical Carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 68Ga-R8760 Dose Selection (Part 1) (Other)
  Interventions: Drug: 68Ga-R8760 injection at pre-defined dose levels
- 68Ga-R8760 Expansion Cohort (Part 2) (Other)
  Interventions: Drug: 68Ga-R8760 injection

INTERVENTIONS:
Drug: 68Ga-R8760 injection at pre-defined dose levels — PET/CT imaging at predefined timepoints
  Arms: 68Ga-R8760 Dose Selection (Part 1)
Drug: 68Ga-R8760 injection — PET/CT imaging at a single timepoint
  Arms: 68Ga-R8760 Expansion Cohort (Part 2)

SUMMARY:
A Phase 1 Safety and Dosimetry Study of 68Ga-R8760 in Patients with Adrenocortical Carcinoma and Healthy Volunteers

ELIGIBILITY:
Adrenocortical Carcinoma Subjects

Inclusion Criteria:

1. Pathologically or clinically confirmed ACC.
2. Newly diagnosed or recurrent/relapsed ACC with at least 1 measurable target lesion per RECIST v1.1 criteria.
3. Male or non-pregnant, non-lactating female subjects age ≥18 years.
4. Female subjects of childbearing potential and male subjects (if sexually active) must agree to use adequate method(s) of effective contraception during their participation in the study.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2.
6. Adequate hepatic function as defined below:

   1. Serum alanine aminotransaminase (ALT)/ aspartate aminotransaminase (AST) ≤3 × upper limit of normal (ULN) or ≤5 × ULN if liver metastases are present or received prior mitotane therapy, and
   2. Serum bilirubin - total ≤1.5 × ULN (unless due to Gilbert's syndrome or hemolysis in which case total ≤3.0 × ULN).
7. Adequate renal function as measured by creatinine clearance calculated by the Cockcroft-Gault formula (≥60 mL/minute).
8. Able to understand and willing to sign a written informed consent form.

Exclusion Criteria:

1. Administered a radionuclide within a period of time corresponding to less than 10 physical half-lives of the radionuclide prior to study Day 1.
2. Radiotherapy ≤14 days prior to study Day 1.
3. Major surgery ≤21 days prior to study Day 1 or has not recovered from adverse effects of such procedure.
4. Severe or unstable medical condition, such as congestive heart failure (New York Heart Association [NYHA] Class III or IV), ischemic heart disease, uncontrolled hypertension, uncontrolled diabetes mellitus, as well as an uncontrolled cardiac arrhythmia requiring medication (≥Grade 2, according to NCI-CTCAE Version 5.0), myocardial infarction within 6 months prior to starting study drug, or any other significant or unstable concurrent cardiac illness. Note: Stable chronic atrial fibrillation is allowed.
5. Congenital long QT syndrome or corrected QT interval by Fridericia (QTcF) interval >450 msec (males) or >470 msec (females).
6. History of cerebrovascular accident within 6 months or that resulted in ongoing neurologic instability.
7. History of other previous or concurrent cancer that would interfere with the determination of safety.
8. Major active infection requiring antibiotics.
9. Known active human immunodeficiency virus infection or active infection with Hepatitis B or C.
10. Acute illness within 14 days prior to study Day 1unless mild in severity, as assessed by the Investigator.
11. Any other condition that in the opinion of the Investigator would place the subject at an unacceptable risk or cause the subject to be unlikely to fully participate or comply with study procedures.

Healthy Volunteers

Inclusion Criteria:

1. Healthy male or non-pregnant, non-lactating female subjects aged between 18 and 59 years (inclusive).
2. Female subjects of childbearing potential and male subjects (if sexually active) must agree to use adequate method(s) of effective contraception during their participation in the study.
3. Body mass index between 18.0 and 32.0 kg/m2 (inclusive).
4. Adequate renal function as measured by creatinine clearance calculated at ≥60 mL/minute by the Cockcroft-Gault formula.
5. Able to understand and willing to sign a written informed consent form.

Exclusion Criteria:

1. Prior unilateral or bilateral adrenalectomy.
2. Mental or legal incapacitation.
3. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
4. Subjects diagnosed with adrenal disease, including Cushing's syndrome, adrenal insufficiency, or congenital adrenal hyperplasia.
5. Glucocorticoid steroid use (including topical) within 4 weeks prior to study Day 1 (inhaled steroids are allowed).
6. Active or recent (within 30 days of screening) infection or history of recurrent chronic infections with underlying condition that may predispose one to infections.
7. Resting pulse rate ≥100 or <40 beats per minute at screening. If abnormal, a repeat measurement will be conducted to confirm.
8. Systolic blood pressure >160 or <90 mmHg or diastolic blood pressure >90 or <50 mmHg, unless judged by the Investigator to have no clinical significance.
9. Participation in a clinical study involving administration of an investigational drug in the past 30 days or 5 half-lives (whichever is longer) prior to study Day 1.
10. Administered a radionuclide within a period of time corresponding to less than 10 physical half-lives of the radionuclide prior to study Day 1.
11. Donation of blood or significant blood loss within 3 months prior to screening, donation of plasma within 2 weeks prior to screening, or donation of platelets within 6 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events characterized overall and by type, frequency, seriousness, relationship to study drug, timing and severity graded according to the NCI-CTCAE v5.0; absolute values and changes in clinical laboratory parameters | 7 days
Absorbed dose coefficients (milliGray [mGy]/megabecquerel [MBq]) in organs | 1 day
The effective dose (milliSievert [mSv]/MBq) | 1 day

SECONDARY OUTCOMES:
Number and location of tumors identified by 68Ga-R8760 PET/CT and by anatomic images | 1 day
Maximum standard uptake value (SUVmax) of each tumor and of source organ | 1 day
Ratio of the tumor SUV over reference region SUV | 1 day
Area under the plasma concentration versus time curse (AUC) | 1 day
Maximum plasma concentration (Cmax) | 1 day
Half-life (T1/2) of 68Ga-R8760 | 1 day

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan Nuclear Medicine, Ann Arbor, Michigan
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No